CLINICAL TRIAL: NCT01070615
Title: A Study to Evaluate the Long-Term Tolerability and Safety of Oral Prucalopride Administered to Patients With Chronic Constipation
Brief Title: Study to Evaluate Long-Term Tolerability and Safety of Oral Prucalopride in Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRU-INT-10
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prucalopride

SUMMARY:
Objectives: Evaluation of the clinical long-term safety, tolerability, patient satisfaction, pharmacokinetics and pattern of use of oral prucalopride tablets given in doses up to 4 mg once daily to patients with chronic constipation

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breast-feeding female outpatients of at least 18 years of age
2. Patient had completed the entire treatment period of the PRU-INT-6 study or the PRU-INT-12 study .

Exclusion Criteria:

1. Patients with impaired renal function
2. Patients with clinically significant abnormalities of haematology, urinalysis, or blood chemistry.
3. Females of child-bearing potential without adequate contraceptive protection during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 1998-06; Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van Outryve, MD, Principal Investigator — University Hospital Antwerp, Edegem, Belgium
Locations (1):
- University Hospital Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] Camilleri M, Van Outryve MJ, Beyens G, Kerstens R, Robinson P, Vandeplassche L. Clinical trial: the efficacy of open-label prucalopride treatment in patients with chronic constipation - follow-up of patients from the pivotal studies. Aliment Pharmacol Ther. 2010 Nov;32(9):1113-23. doi: 10.1111/j.1365-2036.2010.04455.x. Epub 2010 Sep 16. PMID 21039673